CLINICAL TRIAL: NCT04034043
Title: Retrospective Study About Cementless Total Hip Arthroplasty With Ceramic-on-ceramic Bearing Surfaces for Post-traumatic Hip Osteoarthritis After Acetabular Fracture: Long-term Results (ATP)
Brief Title: Ceramic-on-ceramic THA for Post-traumatic Hip Osteoarthritis After Acetabular Fracture
Acronym: APT
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 383/2019/OSS/IOR
Record Dates: First submitted 2019-07-16; First posted 2019-07-26 (Actual); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-07

CONDITIONS: Hip Osteoarthritis; Post-traumatic Osteoarthritis
Keywords: ceramic-on-ceramic; total hip arthroplasty; acetabular fracture; post-traumatic hip osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ceramic-on-ceramic total hip arthroplasty — ceramic-on-ceramic, cementless total hip arthroplasty for post-traumatic hip osteoarthritis.

SUMMARY:
A retrospective consecutive population of patients treated with cementless total hip arthroplasty with ceramic-on-ceramic bearing surfaces due to post-traumatic osteoarthritis due to acetabular fractures will be selected. The aim of this retrospective study is to evaluate the long-term clinical and radiographic results of this implant in such a specific cohort. The secondary aim of the sudy is to provide the complication rate and the failure rate of the cohort. A descriptive analysis of the failures will be provided as well.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) is the recommended treatment to restore functionality and control pain in post-traumatic hip osteoarthritis due to acetabular fractures. However, THA in post-traumatic osteoarthritis following acetabular fractures is a complex procedure and it is burdened with occasional failures. Modest long-term outcomes have been reported, generally lower than conventional THAs performed due to osteonecrosis or primary osteoarthritis: 10-year clinical results are usually good but not excellent (average Harris Hip score: 88), 10-year revision rate is between 15% and 26%. In review study about the complications of post-traumatic THAs, 30% of ossifications, 4.4% of dislocations, 5.6% of infections, and 2.1% of neurovascular lesions were reported: all the percentages were higher than in primary conventional THAs.

The most critical issues are related to the young age of the patients, to the anatomical changes affecting the periarticular tissues, to the presence of hardware and to the greater exposure to septic complications. All these factors may prevent the surgeon to achieve a good cup positioning and a satisfying outcome. However a correct surgical technique, associated with meticulous pre-operative planning and the use of low-wear implants can improve the clinical result and the long term survival rates.

However, the literature about mid-to-long-term studies about post-traumatic THAs is scarce (currently 5 with an average follow-up of at least 5 years). Furthermore, these studies often include outdated implants, positioned with invasive surgical techniques and with removal of all previous hardware. Therefore, a long-term study (minimum 10-year follow-up) involving more recent implants, with modern articular couplings demonstrating low wear (such as ceramic-on-ceramic), and performed with minimally invasive technique and pre-operative CT-guided planning, would be desirable.

The aim of this study is to describe the survival rates and the long-term clinical and radiological outcome (minimum 10-year follow-up) of cementless THAs, with ceramic-on-ceramic couplings, performed with minimally-invasive technique and CT guided pre-operative planning, in post-traumatic osteoarthritis due to acetabular fractures

ELIGIBILITY:
Inclusion Criteria:

* symptomatic, post-traumatic hip osteoarthritis due to acetabular fracture
* consecutive population with a minimum follow-up of 10 years
* cementless total hip arthroplasty with ceramic-on-ceramic bearing surfaces
* pre-operative planning using CT
* complete clinical and radiographic assessment

Exclusion Criteria:

* other type of hip osteoarthritis
* other type of implants
* inadequate pre-operative planning (eg: no CT)
* incomplete assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: retrospective, consecutive population treated with a cementless total hip arthroplasty with ceramic-on-ceramic bearing surfaces for post-traumatic hip osteoarthritis due to acetabular fracture. A minimum follow-up of 10 years was mandatory.
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-07-19 (Actual); Study Completion 2019-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Traina, MD, Study Chair — IRCCS Istituto Ortopedico Rizzoli
Locations (1):
- IRCSS Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bellabarba C, Berger RA, Bentley CD, Quigley LR, Jacobs JJ, Rosenberg AG, Sheinkop MB, Galante JO. Cementless acetabular reconstruction after acetabular fracture. J Bone Joint Surg Am. 2001 Jun;83(6):868-76. doi: 10.2106/00004623-200106000-00008. PMID 11407795
- [Result] Makridis KG, Obakponovwe O, Bobak P, Giannoudis PV. Total hip arthroplasty after acetabular fracture: incidence of complications, reoperation rates and functional outcomes: evidence today. J Arthroplasty. 2014 Oct;29(10):1983-90. doi: 10.1016/j.arth.2014.06.001. Epub 2014 Jun 12. PMID 25034883
- [Result] Weber M, Berry DJ, Harmsen WS. Total hip arthroplasty after operative treatment of an acetabular fracture. J Bone Joint Surg Am. 1998 Sep;80(9):1295-305. doi: 10.2106/00004623-199809000-00008. PMID 9759814
- [Result] Berry DJ. Total hip arthroplasty following acetabular fracture. Orthopedics. 1999 Sep;22(9):837-9. doi: 10.3928/0147-7447-19990901-14. No abstract available. PMID 10507340
- [Result] Ranawat A, Zelken J, Helfet D, Buly R. Total hip arthroplasty for posttraumatic arthritis after acetabular fracture. J Arthroplasty. 2009 Aug;24(5):759-67. doi: 10.1016/j.arth.2008.04.004. Epub 2008 Jun 4. PMID 18534534
- [Result] Lai O, Yang J, Shen B, Zhou Z, Kang P, Pei F. Midterm results of uncemented acetabular reconstruction for posttraumatic arthritis secondary to acetabular fracture. J Arthroplasty. 2011 Oct;26(7):1008-13. doi: 10.1016/j.arth.2011.02.026. Epub 2011 Apr 6. PMID 21474274

RESULTS

PARTICIPANT FLOW:
Groups:
- THA Post Acetabular Fractures: Ceramic-on-ceramic THA for Post-traumatic Hip Osteoarthritis After Acetabular Fracture with a minimum follow-up of 10 years
Period: Overall Study
Arm/Group | THA Post Acetabular Fractures
Started | 68
Completed | 68
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | THA Post Acetabular Fractures
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 68
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 68
percentages of patients treated operatively [Count of Participants; unit: Participants] | 50

OUTCOME MEASURES:

1. Primary Outcome: Survival Rates of the Hip Implants
Description: Kaplan Meier curve with 95% confidence intervals
Time Frame: 10 years-18 years
Measure: Mean (95% Confidence Interval); unit: percentage of non-revised implants
Arm/Group | THA Post Acetabular Fractures
Number analyzed (Participants) | 68
percentage of non-revised implants | 96.3 [86.1 to 99.1]

2. Primary Outcome: Clinical Outcomes of the Hip Implants
Description: HHS score (Harris Hip Score). Total scale: 0-100. Best performance: 100
Time Frame: 10 years-18 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THA Post Acetabular Fractures
Number analyzed (Participants) | 68
score on a scale | 88.4 (11.6)

3. Primary Outcome: Clinical Outcomes of the Hip Implants
Description: WOMAC score (Western Ontario and McMaster Universities Osteoarthritis Index). Total scale: 0-96. Best performance: 96
Time Frame: 10 years -18 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | THA Post Acetabular Fractures
Number analyzed (Participants) | 68
score on a scale | 84.3 (9.6)

4. Primary Outcome: Percentage of Patients With Adequate Radiographic Cup Osseointegration
Description: Percentage of patients with a good osseointegration defined by the criteria described by Moore et al. Measurement technique: qualitative visual assessment of 5 binary parameters (yes/no): radial trabeculae, stress shielding, superolateral buttress, inferomedial buttress, absence of radiolucent lines. Adequate osseointegration: at least 3 parameters are present. Total scale: 0%-100%. Best performance (every patient has adequate osseointegration at 10 years): 100
Time Frame: 10 years-18 years
Measure: Count of Participants; unit: Participants
Arm/Group | THA Post Acetabular Fractures
Number analyzed (Participants) | 68
Participants | 68

ADVERSE EVENTS:
Time Frame: 10 years-18 years
Arm/Group | THA Post Acetabular Fractures
All-Cause Mortality (participants affected / at risk) | 0/68
Serious Adverse Events (participants affected / at risk) | 8/68
Other Adverse Events (participants affected / at risk) | 2/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THA Post Acetabular Fractures (N=68)
modular neck failure (Musculoskeletal and connective tissue disorders) | 4 (4)
periprosthetic fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Aseptic loosening of the stem (Musculoskeletal and connective tissue disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | THA Post Acetabular Fractures (N=60)
Dislocation not requiring revision surgery (Musculoskeletal and connective tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT04034043/Prot_SAP_000.pdf